CLINICAL TRIAL: NCT07044375
Title: Going Places: A Multi-level Intervention to Improve Youth Transportation Efficacy and Physical Activity
Acronym: Going Places
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Durham Parks and Recreation (Durham, NC) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00106083
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Physical Activity; Cardiometabolic Risk Factors; Cardiometabolic Health Indicators; Self-Efficacy
Keywords: Program planning and implementation; Community youth organizations; Community-based physical activity; Transportation self-efficacy; Cardiometabolic health; Physical activity; Parks and Recreation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Going Places (Other): Teens enrolled in the MyDurham park-based afterschool program will receive the Going Places youth transportation intervention.
  Interventions: Behavioral: Going Places

INTERVENTIONS:
Behavioral: Going Places — Going Places is a community driven intervention to increase transportation self-efficacy among low-income youth, enabling access to community-based programs that promote physical activity and improve long term cardiometabolic health. The intervention incorporates a multi-level approach that includes 1) workshops on navigating local transportation systems; 2) field trips and participatory assets mapping activities; and 3) youth transportation advocacy.

SUMMARY:
Going Places is a community driven intervention to increase transportation self-efficacy among low-income youth, enabling access to community-based programs that promote physical activity and improve long term cardiometabolic health. Going Places was co-developed under the joint leadership of Duke and Durham Parks and Recreation (DPR). Going Places is pilot tested and fully functional. The intervention incorporates a multi-level approach that includes 1) workshops on navigating local transportation systems; 2) field trips and participatory assets mapping activities; and 3) youth transportation advocacy.

DETAILED DESCRIPTION:
Going Places is a multilevel transportation self-efficacy intervention designed to increase physical activity (PA) among under resourced youth and improve their cardiometabolic health. Going Places is informed by the Socioecological Framework and Bandura's Self-efficacy Theory and includes the following components: weekly workshops on navigating transportation systems (individual level), community field trips and participatory mapping activities (recreation center level), and local transportation advocacy (environment level). Going Places was codeveloped under the joint leadership of Duke University and Durham Parks and Recreation (DPR; Durham, NC).

Going Places is offered to individual youth as part of DPR's no-cost adolescent afterschool program for youths aged 13 to 19 years. Going Places provides weekly workshops co-led by Duke and DPR that aimed to promote transportation self-efficacy (e.g., how to use local transportation systems, including biking and walking path trail maps, acquiring a free bus pass, using the bus and rail system, pedestrian and biking safety). Workshops also include engaging in active games and recreation.

Monthly field trips organized with the recreation center provide opportunities for youth to navigate transportation systems and engage in PA, primarily in outdoor settings. Youth also participate in a series of participatory mapping exercises to identify safe routes to reach neighborhood sites for active recreation.

The intervention's environmental components focus on promoting access to transportation and PA for youths. The Going Places study team, youth participants, and the program's Steering Committee collaborate with local organizations that oversee recreation and transportation programs and policy in Durham. These organizations are involved in ongoing advocacy to promote safe, affordable, and sustainable transportation and recreation, including park renovation and restoration projects, public mural contests, and social activism (web; social media).

ELIGIBILITY:
Inclusion Criteria:

* Age 12-18 years
* 18 years or older and has a family member who or has enrolled in Durham Parks and Recreation programs
* Enrolled in the MyDurham teen park-based afterschool program in Durham, NC
* Reads, writes and speaks English
* Durham Parks and Recreation Staff

Exclusion Criteria:

* Age <12 years or >18 years
* Not enrolled in the MyDurham teen park-based afterschool program in Durham, NC

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical Activity as measured by number of steps per day | Baseline and 4 months
  Youth participants were provided with Garmin accelerometers at baseline and 4 months to monitor step data over 7 consecutive days. Wrist-worn accelerometry (versus waist worn) was chosen to maximize compliance. A threshold of 11,500 or more steps per day was used to evaluate whether participants met daily steps goals.
Transportation Self-Efficacy as measured by the Teen Environment and Neighborhood (TEAN) scale | Baseline and 4 months
  The primary measure of youth transportation self-efficacy measured at baseline and 4 months will be the Teen Environment and Neighborhood (TEAN) scale, measured via surveys collected during regular youth program hours.
Transportation Self-Efficacy as measured by the Youth Living in Active Neighborhoods scale | Baseline and 4 months
  The Youth Living in Active Neighborhoods scale is a 67-item questionnaire that assesses youth perceptions of neighborhood design features related to physical activity. A higher score indicates greater neighborhood walkability.
Transportation Self-Efficacy as measured by Physical Activity Neighborhood Environment Scale (PANES) | Baseline and 4 months
  The PANES is used to assess the environmental factors for walking and bicycling in the participant's neighborhood. The score is calculated as a mean of items 1 through 17 and has a range of 1 to 4, with higher values indicating greater environmental support for physical activity.

SECONDARY OUTCOMES:
Moderate-to-Vigorous Physical Activity (MVPA) time per day | Baseline and 4 months
  Data will be summarized to compute participant-level moderate-to-vigorous PA corresponding to each time point. Wrist worn accelerometry (versus waist worn) was chosen to maximize compliance.
Total Physical Activity (PA) time per day | Baseline and 4 months
  Total PA includes all non-sedentary time. Data will be summarized to compute participant-level total PA per day corresponding to each time point. Wrist worn accelerometry (versus waist worn) was chosen to maximize compliance.
Systolic Blood Pressure (SBP) | Baseline and 4 months
  A total of three SBP measurements will be taken successively with 1-min in between each measure. For analysis, the first value will be dropped, and the subsequent two will be averaged.
Diastolic Blood Pressure (DBP) | Baseline and 4 months
  A total of three DBP measurements will be taken successively with 1-min in between each measure. For analysis, the first value will be dropped, and the subsequent two will be averaged.

CONTACTS AND LOCATIONS:
Overall Officials: Emily D'Agostino, DPH, MS, MEd, MA, Principal Investigator — Duke University
Locations (1):
- Durham Parks and Recreation, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller HN, Berger MB, Askew S, Trefney E, Tyson C, Svetkey L, Bennett GG, Steinberg DM. Implementation of an At-home Blood Pressure Measurement Protocol in a Hypertension Management Clinical Trial During the COVID-19 Pandemic. J Cardiovasc Nurs. 2022 Sep-Oct 01;37(5):475-481. doi: 10.1097/JCN.0000000000000927. Epub 2022 Apr 23. PMID 35467561
- [Background] Urbina E, Alpert B, Flynn J, Hayman L, Harshfield GA, Jacobson M, Mahoney L, McCrindle B, Mietus-Snyder M, Steinberger J, Daniels S; American Heart Association Atherosclerosis, Hypertension, and Obesity in Youth Committee. Ambulatory blood pressure monitoring in children and adolescents: recommendations for standard assessment: a scientific statement from the American Heart Association Atherosclerosis, Hypertension, and Obesity in Youth Committee of the council on cardiovascular disease in the young and the council for high blood pressure research. Hypertension. 2008 Sep;52(3):433-51. doi: 10.1161/HYPERTENSIONAHA.108.190329. Epub 2008 Aug 4. No abstract available. PMID 18678786
- [Background] National High Blood Pressure Education Program Working Group on High Blood Pressure in Children and Adolescents. The fourth report on the diagnosis, evaluation, and treatment of high blood pressure in children and adolescents. Pediatrics. 2004 Aug;114(2 Suppl 4th Report):555-76. No abstract available. PMID 15286277
- [Result] Chung NW, Ostbye T, Jones JM, Smith AL, Zewdie HY, Yuan A, Kumar A, D'Agostino EM. Needs Assessment and Feasibility of a Park-Based Active Transportation Intervention to Promote Youth Physical Activity and Access to Parks and Recreation. Journal of Park and Recreation Administration. 2023 July. DOI:10.18666/JPRA-2023-11830
- [Result] D'Agostino EM, Neshteruk CD, Li T, Davis J, Granados I, Kumar A, Forde J, Hornik CP. Going Places: An Active Transportation Intervention to Increase Youth Physical Activity, Durham, North Carolina, 2023-2024. Am J Public Health. 2025 May;115(5):693-697. doi: 10.2105/AJPH.2025.308012. Epub 2025 Mar 20. PMID 40112267